CLINICAL TRIAL: NCT05989438
Title: Analysis of the Impact of Different Intervention Models on the Neuropsychomotor Development of Premature Infants Based on the ICF Biopsychosocial Model
Brief Title: Different Intervention Models of Premature Infants Based on the ICF Biopsychosocial Model
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fernanda Cechetti, PrematurityICF, Federal University of Health Science of Porto Alegre
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PrematurityICF
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Prematurity
Keywords: Prematurity; Physiotherapy; CIF; Child development; Early Intervention
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premature that the family receives only orientation. (Active Comparator): The orientations will happen once a month via telephone, and once a week a reminder will be sent. Follow-up will occur from 4 to 12 corrected months.
  Interventions: Other: Orientations for families
- Premature who receive intervention by a specialized professional more orientation for the family (Active Comparator): The frequency of stimulation by a specialized professional will vary according to the degree of prematurity, from approximately 1 to 8 times per month. The guidelines will take place on the days of the calls. Follow-up will occur from 4 to 12 corrected months.
  Interventions: Other: Professional stimulation more orientations for families.

INTERVENTIONS:
Other: Orientations for families — Guidance for parents will follow the guide/manual prepared by the researchers, in addition to verbal and video guidance. Once a week a reminder will be sent, and once a month researchers will contact you by phone for guidance.
  There will be 3 evaluations with an interval of 4 months. (4 months; 8 months; 12 months) and more one avaliation with an interval of 12 months at 24 months.
  Arms: Premature that the family receives only orientation.
Other: Professional stimulation more orientations for families. — Each session will last approximately 50 minutes, where the stimuli will be performed in: supine position; Ventral Decubitus; Seated; Four supports, kneeling/semi-kneeling and standing.
  If the child no longer uses the posture or it is not an acquisition for the age group in which the baby is, the time will be distributed in order to contemplate the expected acquisitions for the age group in which the baby is. The stimuli will be performed based on the neuropsychomotor development, in order of progression and according to the corrected age of the baby.
  The frequency of consultations may vary due to the different degrees of prematurity, and the stipulated initial frequency will vary between 1-8 times a month.
  The orientations will also be provided to family members during consultations, and families will also perform stimuli at home according to written, verbal and video guidance.
  There will be 3 evaluations with an interval of 4 months. (4 months; 8 months; 12 months).
  Arms: Premature who receive intervention by a specialized professional more orientation for the family

SUMMARY:
Prematurity is an important risk factor for delayed neuropsychomotor development. The main objective of this study is to analyze the impact of different intervention models on the neuropsychomotor development of premature babies based on the ICF biopsychosocial model.

DETAILED DESCRIPTION:
Premature birth is defined as one in which it occurs before 37 completed weeks of gestation. Prematurity is due to different circumstances, and premature babies can be classified according to gestational age as extremely premature, very premature, or moderately to late preterm. Prematurity is one of the main biological risk factors, and that it contributes to the appearance of changes in the neuropsychomotor development of babies, which may compromise their functional capacity. Thus, screening is essential so that families are guided and premature babies receive adequate early intervention through follow-up programs, mainly aimed at functionality. Given this, and to help standardize health approaches, since 2001 with the development of the biopsychosocial model of health, based on the International Classification of Functioning, Disability and Health (ICF), the use of the ICF is recommended in research and in clinical practice. However, although the use of the ICF in interventions is recommended worldwide, and the literature shows a growing increase in the use of the ICF in studies involving children and young people, there is a shortage of studies, especially in what culminates neuropsychomotor development and prematurity. Thus, the main objective of this study is to analyze the impact of different interventional models on the neuropsychomotor development of premature babies based on the biopsychosocial model of the ICF. This is a randomized, uncontrolled clinical trial, participants will be premature babies with corrected age between 4 and 24 months. Parents of babies who meet the proposed inclusion criteria will be invited to allow participation by signing the Free and Informed Consent term.

The study is composed of two large groups: Stimulation plus Orientations Group and Orientations Group. Participants in both groups will follow the same inclusion and exclusion criteria. Regardless of delay in neuropsychomotor development, during and at the end of each of the three assessments, parents or guardians from both groups received verbal guidance. In addition, in the first evaluation, a printed guide with guidelines for stimulating the baby at home will be given to all families, where the guidelines were divided by months, encompassing from 4 to 24 corrected months.

The guidance guide for families was produced by the researchers emphasizing appropriate stimuli for the corrected age. The guide aims to stimulate neuropsychomotor development, in order to give the baby the opportunity to experiment with new skills, through different postures and transfers, and through facilitation, motor, cognitive, auditory, visual and sensory stimuli. The guidelines prioritize rudimentary postures (prone, supine, lateral decubitus, sitting and standing), in addition to stimuli on cognitive, language, visual and auditory aspects. Parents or guardians will be asked to stimulate their children daily, at the time that is most appropriate for the family's routine, strengthening the bond with the baby. Control of the frequency of performing the stimuli at home will be carried out, the control will be carried out by the families themselves by filling in a column in the guide for information on frequency. The researchers will get in touch with the families in the guidance group once a month to guide and clarify possible doubts, while the families in the guidance plus stimulation group, as they will attend more often than once a month, will have the opportunity to clarify doubts directly with the researcher during the consultations. The researchers will also be available to all families in both groups throughout the entire survey over the phone.

Thinking that we can find families with unfavorable socioeconomic conditions and, also, with the intention of standardizing the stimuli, appropriate toys for each age group will be delivered to all families in the two groups, which will be made by the researchers.

All babies in both groups will participate in a follow-up program where assessments will take place in 4 moments with an interval of 4 months between them on the first year of life (tolerating a window of one month and a half), where: initial assessment, time 1 (t1): 4 corrected months; time 2 (t2): 8 corrected months; time 3 (t3) 12 months corrected; on the time 4 (t4) (will be tolerating a window of four months), 24 months corrected for extreme birth babies (< 28 weeks gestational age) and 24 months cronologic for babies ≥ 28 weeks gestational age. There will be four moments of evaluation that will consist of the analysis of:

* Neuropsychomotor development through the Bayley Infant and Toddler Development Scales, third edition (Bayley III);
* Montreal Cognitive Assessment (MoCA).
* Patient identification data through an evaluation questionnaire and initial anamnesis, information from the health booklet and data from the medical record.
* Affordances in the Home Environment through Affordances in the Home Environment for Motor Development - Children's Scale (AHEMD-IS);
* Quality of life through the Pediatric Inventory on Baby Quality of Life (PedsQL®);
* Socioeconomic data through the Socioeconomic Questionnaire of the Brazilian Research Association (ABEP).
* Parents' cognitive assessment through the Montreal Cognitive Assessment (MoCA).

ELIGIBILITY:
Inclusion Criteria:

* 1. Gestational age less than 37 weeks, corrected age between 4 and 12 months (one and a half month window) and at 24 months (four months window)
* Babies from the High Risk Outpatient Clinic of the UCS Clinical Center, registered there;
* Authorization of those responsible for the minor consenting to participation in the study by signing the Free and Informed Consent Form (TCLE).

Exclusion Criteria:

* All those subjects who do not follow the items mentioned above;
* Presenting neurological diseases;
* Presence of acute diseases (eg pneumonia, bronchiolitis, trauma)
* Musculoskeletal alterations;
* Genetic syndromes;
* In genetic investigation;
* Heart diseases with indication for surgical intervention;
* Untreated congenital torticollis;
* Congenital clubfoot;
* Cerebral hemorrhage grade IV
* Those who do not undergo the first and/or last evaluation;
* Incomplete evaluation;
* Convulsive crisis during study period;
* Participants from other intervention programs.

Ages: 4 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-01-11 (Estimated)

PRIMARY OUTCOMES:
Bayley III | 24 months
  The Bayley Scales of Infant and Child Development - 3rd Edition, consist of an instrument applied individually to assess the development of children between 1 and 42 months of age and are widely used in research and clinical practice to assess child development. They enable early diagnosis of developmental delays, providing information for planning and intervention. It can be used, for example, to evaluate children, typical, atypical, term or premature. The Bayley-III provides the examiner with the ability to adjust scores for prematurity up to 24 months, which is one of the most notable features of the scale. The adjustment corrects the child's age to his expected chronological age if he had been born at term.
  Currently in its third edition, Bayley III presents five distinct subtests for assessing child development in the areas of cognition, language, motor, socio-emotional and adaptive behavior.

SECONDARY OUTCOMES:
Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS) | 24 months
  The AHEMD-IS is a validated and reliable instrument for the assessment of infants aged 3 to 18 months. The instrument consists of 35 items divided into 4 dimensions (Physical Space, Variety of Stimulation, Fine Motor Toys and Gross Motor Toys) and a total score that can be categorized into 4 descriptions of domestic motor affordances (scoring system): Insufficient, Moderately Adequate, Adequate and Excellent. The results suggest that this tool can be a useful tool to measure the quantity and quality of affordances in the home environment that favor children's motor development. Researchers will be able to use this instrument to explain this important contributor to children's motor development, as well as for evaluation and intervention recommendations, in addition to advising parents on household activities.
Pediatric Baby Quality of Life Inventory (PedsQL@) | 24 months
  When considering that gains in quality of life in relation to an intervention process are desired outcomes from the perspective of favoring a good health condition, according to the BPS model of the ICF, the Pediatric Inventory on the quality of life of babies presents validity and reliability to be used both in healthy children and those with illnesses or atypical development. It presents versions according to age and health condition. For babies, it presents a version for 1-12 months and another for 13-24 months and is carried out by interviewing parents and/or caregivers. It allows the assessment of quality of life in relation to physical capacity, physical symptoms, emotional aspects, social interaction, cognition and a total score. In cases of specific health conditions or older children, there are specific forms.
Socioeconomic Questionnaire for Brazil | 24 months
  The Socioeconomic Questionnaire for Brazil (ABEP) is a questionnaire used for socioeconomic definition. He reviews all items of appliances that are working, including those that are in storage, or if they are not working, but the family considers fixing or replacing them in 6 months. The points system is composed of the variables: Bathrooms, domestic servants, cars, microcomputer, dishwasher, refrigerator, freezer, washing machine, microwave, motorcycle, clothes dryer (scoring according to the quantity: 0, 1, 2 , 3, 4 or more).
  In addition, I evaluate the level of education of the head of the family:
  * Illiterate / Incomplete elementary school: 0 points
  * Complete Elementary I / Incomplete Elementary II: 1 point
  * Complete Elementary II / Incomplete High School: 2 points
  * Incomplete Middle School / Incomplete Higher Education: 4 points
  * Higher education: 7 points And this instrument also analyzes the conditions of public services for the items: piped
Montreal Cognitive Assessment-MoCA | 24 months
  The MoCA (Montreal Cognitive Assessment) test will be used in this study as a tool for the cognitive assessment of parents, aiming to identify possible changes in cognitive functions, even if subtle. It is a validated and widely used tool in the screening of mild cognitive impairment, offering a comprehensive analysis of skills such as memory, attention, language, executive function and orientation. The application of the MoCA will allow a standardized and objective assessment of the cognitive performance of the participants, contributing to a better understanding of the cognitive profile of the parents in the study sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre (UFCSPA), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No